CLINICAL TRIAL: NCT00758186
Title: Endoscopic Stenting and Elective Surgery Versus Emergency Surgery for Left-sided Malignant Colonic Obstruction: A Prospective Randomized Trial.
Brief Title: Randomized Trial of Colonic Stents as a Bridge to Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Colonic-Stenting-001
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Colorectal Cancer; Intestinal Obstruction
Keywords: Colorectal cancer; Endoscopic stent; Intestinal obstruction; Laparoscopy
MeSH Terms: conditions — Colorectal Neoplasms; Intestinal Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Colonic-stenting (Experimental): Colonic-stenting and elective surgery: Emergency endoscopic colonic stenting followed by elective surgery at a later date for acute left-sided malignant colonic obstruction.
  Interventions: Procedure: Emergency endoscopic colonic stenting
- Emergency surgery (Active Comparator): Emergency surgery: Patients underwent emergency surgery for acute left-sided malignant colonic obstruction.
  Interventions: Procedure: Emergency surgery

INTERVENTIONS:
Procedure: Emergency endoscopic colonic stenting — Colonic-stenting and elective surgery: Emergency endoscopic colonic stenting followed by elective surgery at a later date for acute left-sided malignant colonic obstruction. Patients who had successful stenting were discharged and re-admitted for elective surgery. Patients in whom stenting was unsuccessful underwent emergency surgery. The choice of surgery performed was up to the individual consultant colorectal surgeon.
  Arms: Colonic-stenting
Procedure: Emergency surgery — Patients underwent emergency surgery for acute left-sided malignant colonic obstruction. The choice of surgery performed was up to the individual consultant colorectal surgeon. Surgery included primary resection with or without defunctioning stoma and palliative diverting stoma only.
  Arms: Emergency surgery

SUMMARY:
The objective of this randomized controlled trial was to evaluate the role colonic self-expanding metal stent (SEMS) placement as a bridge to surgery in patients with acute malignant left-sided colonic obstruction. The study was designed to test the hypothesis that SEMS placement could be effectively and safely used in this group of patients to relieve colonic obstruction thereby allowing safe recovery and medical stabilization before proceeding to elective surgery

ELIGIBILITY:
Inclusion Criteria:

* Acute intestinal obstruction secondary to left-sided colonic cancer

Exclusion Criteria:

* Distal rectal cancers
* Patients with signs of peritonitis suggestive of bowel perforation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-10; Primary Completion 2008-02 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
The primary endpoint was postoperative complication rates. | 30 days

SECONDARY OUTCOMES:
Secondary outcomes evaluated included type of surgery performed, bowel preservation, presence of a stoma, postoperative bowel function, length of hospital stay, and hospitalization costs. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Kok-Sun Ho, FRCSEd, Principal Investigator — Department of Colorectal Surgery, Singapore General Hospital
Locations (1):
- Department of Colorectal Surgery, Singapore General Hospital, Singapore, Singapore

REFERENCES:
- [Background] Lim JF, Tang CL, Seow-Choen F, Heah SM. Prospective, randomized trial comparing intraoperative colonic irrigation with manual decompression only for obstructed left-sided colorectal cancer. Dis Colon Rectum. 2005 Feb;48(2):205-9. doi: 10.1007/s10350-004-0803-9. PMID 15714241
- [Background] Saida Y, Sumiyama Y, Nagao J, Uramatsu M. Long-term prognosis of preoperative "bridge to surgery" expandable metallic stent insertion for obstructive colorectal cancer: comparison with emergency operation. Dis Colon Rectum. 2003 Oct;46(10 Suppl):S44-9. doi: 10.1097/01.DCR.0000087483.63718.A2. PMID 14530657
- [Background] Martinez-Santos C, Lobato RF, Fradejas JM, Pinto I, Ortega-Deballon P, Moreno-Azcoita M. Self-expandable stent before elective surgery vs. emergency surgery for the treatment of malignant colorectal obstructions: comparison of primary anastomosis and morbidity rates. Dis Colon Rectum. 2002 Mar;45(3):401-6. doi: 10.1007/s10350-004-6190-4. PMID 12068202
- [Background] Khot UP, Lang AW, Murali K, Parker MC. Systematic review of the efficacy and safety of colorectal stents. Br J Surg. 2002 Sep;89(9):1096-102. doi: 10.1046/j.1365-2168.2002.02148.x. PMID 12190673